CLINICAL TRIAL: NCT02435212
Title: A Randomized, Open-label, Multicenter, Two Arm, Phase II Study to Evaluate Treatment Compliance, Efficacy and Safety of an Improved Deferasirox Formulation (Granules) in Pediatric Patients With Iron Overload
Brief Title: Study to Evaluate Treatment Compliance, Efficacy and Safety of an Improved Deferasirox Formulation (Granules) in Pediatric Patients (2-<18 Years Old) With Iron Overload
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670F2202; 2013-004739-55 (EudraCT Number)
Record Dates: First submitted 2015-03-17; First posted 2015-05-06 (Estimated); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Transfusion-dependent Anemia
Keywords: New formulation; deferasirox; chelation; iron overload; compliance; satisfaction; palatability; PRO; PK; safety; PK/PD; ICL670
MeSH Terms: conditions — Iron Overload; Patient Compliance; Personal Satisfaction | interventions — Deferasirox

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DFX DT (Active Comparator): Participants will be administered deferasirox dispersible tablets orally once daily based on body weight for 48 weeks.
  Interventions: Drug: Deferasirox DT formulation
- DFX Granule (Experimental): Participants will be administered deferasirox granules orally once daily in the form of stick packs based on body weight for 48 weeks.
  Interventions: Drug: Deferasirox granule formulation

INTERVENTIONS:
Drug: Deferasirox granule formulation — Deferasirox granules will be provided as stick packs containing 90 mg, 180 mg and 360 mg granules for oral use and will be administered based on body weight.
  Other Names: ICL670
  Arms: DFX Granule
Drug: Deferasirox DT formulation — Deferasirox DT will be provided as 125 mg, 250 mg and 500 mg dispersible tablets for oral use and will be administered based on body weight.
  Other Names: ICL670
  Arms: DFX DT

SUMMARY:
This was a randomized, open-label, multicenter, two arm, phase II study to evaluate treatment compliance and change in serum ferritin of a deferasirox granule formulation and a deferasirox dispersible tablet (DT) formulation in children and adolescents aged ≥ 2 and < 18 years at enrolment with any transfusion-dependent anemia requiring chelation therapy due to iron overload, to demonstrate the effect of improved compliance on iron burden.

Randomization was stratified by age groups (2 to <10 years, 10 to <18 years) and prior iron chelation therapy (Yes/ No). There were two study phases which include a 1 year core phase where participants were randomized to a 48 week treatment period to either Deferasirox DT or granules, and an optional extension phase where all participants received the granules up to 5 years. Participants who demonstrated benefit to granules or DT in the core phase, and/or expressed the wish to continue in the optional extension phase on granules, were offered this possibility until there was local access to the new formulation (granules or film-coated tablet (FCT)) or up to 5 years, whichever occurred first.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent/assent before any study-specific procedures. Consent will be obtained from parent(s) or legal guardians. Investigators will also obtain assent of patients according to local guidelines.
* Male and female children and adolescents aged ≥ 2 and < 18 years. [France: Male and female children and adolescent aged ≥ 2 and < 18 years old, however children aged ≥ 2 and ≤ 6years can be enrolled only when deferoxamine treatment is contraindicated or inadequate in these patients as per investigator decision. Applicable to core phase only. Once in the core phase patients can turn 18 years and still be considered eligible, also for participation in the optional extension phase.
* Any transfusion-dependent anemia associated with iron overload requiring iron chelation therapy and with a history of transfusion of approximately 20 PRBC units and a treatment goal to reduce iron burden (300mL PRBC = 1 unit in adults whereas 4 ml/kg PRBC is considered 1 unit for children).
* Serum ferritin > 1000 ng/mL, measured at screening Visit 1 and screening Visit 2 (the mean value will be used for eligibility criteria).
* Patient has to have participated and completed the 48 weeks core phase treatment as per protocol (For optional extension phase eligibility only).

Exclusion Criteria:

* Creatinine clearance below the contraindication limit in the locally approved prescribing information (using Schwartz formula) at screening visit 1 or screening visit 2.
* Serum creatinine > 1.5 xULN at screening measured at screening Visit 1 and or screening Visit 2
* ALT and/or AST > 3.0 x ULN at screening visit 1 or screening visit 2..
* Liver disease with severity of Child-Pugh class B or C.
* Significant proteinuria as indicated by a urinary protein/creatinine ratio > 0.5 mg/mg in a second morning urine sample at screening Visit 1 or screening Visit 2.
* Patients with significant impaired gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral deferasirox (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome or small bowel resection).
* Direct (conjugated) bilirubin >2 x ULN at screening visit 1 or screening visit 2.
* Local access to new formulation (granules or FCT) is available (For optional extension phase eligibility only).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 224 (Actual)
Dates: Start 2015-10-21 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2024-01-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (42):
- United States (13):
  - Novartis Investigative Site, Oakland, California
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Chicago, Illinois
  - Novartis Investigative Site, New York, New York
  - Weill Cornell Medical College SC -, New York, New York
  - Childrens Hospital at Montefiore, The Bronx, New York
  - Novartis Investigative Site, The Bronx, New York
  - Childrens Hospital of Philadelphia Onc. Dept, Philadelphia, Pennsylvania
  - Novartis Investigative Site, Philadelphia, Pennsylvania
  - Medical Uni of South Carolina Medical Uni of South Carolina, Charleston, South Carolina
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Memphis, Tennessee
  - St. Jude Children's Research Hospital Memphis St Jude, Memphis, Tennessee
- Belgium (2):
  - Novartis Investigative Site, Edegem, Antwerpen
  - Novartis Investigative Site, Brussels
- Bulgaria (3):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Varna
- Novartis Investigative Site, Alexandria, Egypt
- France (2):
  - Novartis Investigative Site, Créteil
  - Novartis Investigative Site, Paris
- Novartis Investigative Site, Debrecen, Hungary
- Novartis Investigative Site, Kolkata, West Bengal, India
- Italy (3):
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Palermo, PA
  - Novartis Investigative Site, Napoli
- Novartis Investigative Site, Hazmiyeh, Beyrouth, Lebanon
- Malaysia (4):
  - Novartis Investigative Site, Ipoh, Perak
  - Novartis Investigative Site, Kuching, Sarawak
  - Novartis Investigative Site, Kuala Lumpur
  - Novartis Investigative Site, Pulau Pinang
- Novartis Investigative Site, Muscat, Oman
- Novartis Investigative Site, Panama City, Republica de Panama, Panama
- Philippines (2):
  - Novartis Investigative Site, Quezon
  - Novartis Investigative Site, Quezon City
- Novartis Investigative Site, Moscow, Russia
- Thailand (2):
  - Novartis Investigative Site, Bangkok Noi, Bangkok
  - Novartis Investigative Site, Muang, Chiangmai
- Novartis Investigative Site, Tunis, Tunisia
- Turkey (Türkiye) (3):
  - Novartis Investigative Site, Adana
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Izmir

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After enrollment, participants previously treated with iron chelation therapy (ICT) underwent a 5-day chelation washout period prior to the commencement of the 48-week treatment (Core phase).
Groups:
- DFX DT: Participants received deferasirox (DFX) dispersible tablets (DT) orally once daily based on body weight for 48 weeks in the Core phase. The starting dose was 20mg/kg/day which was then adjusted based on tolerability, safety and efficacy considerations. After the Core phase, participants could enter the Optional Extension phase and cross over to DFX granules administered orally once daily in the form of stick packs for up to 5 years. Participants entering the Optional Extension phase received the equivalent strength-adjusted DFX granules dose corresponding to the last DT dose in the Core phase taking dose adjustment guidelines into account.
- DFX Granule: Participants received deferasirox (DFX) granules orally once daily based on body weight in the form of stick packs for 48 weeks in the Core phase. The starting dose was 14 mg/kg/day which was then adjusted based on tolerability, safety and efficacy considerations. After the Core phase, participants could enter the Optional Extension phase and continued receiving DFX granules at the same dose as was given at the end of the Core phase taking dose adjustment guidelines into account for up to 5 years.
Period: Core Phase
Arm/Group | DFX DT | DFX Granule
Started | 112 | 112
Completed | 87 | 99
Not Completed | 25 | 13
Not completed — Adverse Event | 8 | 5
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Withdrawal by parent/guardian | 9 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Physician Decision | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Lack of Efficacy | 0 | 1
Not completed — Recovery | 1 | 0
Period: Optional Extension Phase
Arm/Group | DFX DT | DFX Granule
Started | 69 | 77
Completed | 42 | 46
Not Completed | 27 | 31
Not completed — Adverse Event | 3 | 9
Not completed — Physician Decision | 6 | 8
Not completed — Withdrawal by parent/guardian | 10 | 7
Not completed — Lack of Efficacy | 2 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Recovery | 1 | 1
Not completed — Death | 1 | 0
Not completed — Technical problems | 2 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) was defined according to the Intent to Treat (ITT) principle, and included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | DFX DT | DFX Granule | Total
Number analyzed (Participants) | 112 | 112 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.8 (3.89) | 5.9 (3.94) | 5.9 (3.90)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 54 | 56 | 110
  Male | 58 | 56 | 114
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 7 | 14
  Not Hispanic or Latino | 104 | 105 | 209
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 38 | 44 | 82
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 57 | 52 | 109
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Overall Compliance Using Stick Pack or Tablet Counts in Iron Chelation Therapy (ICT)-naïve Participants During the Core Phase
Description: Compliance was calculated as the ratio of total count consumed to total count prescribed of deferasirox granule stick packs or dispersible tablets, where total count consumed was derived from cumulative dispensed, returned and lost/wasted counts over 24 weeks of treatment and total count prescribed was derived from cumulative prescribed count over 24 weeks of treatment.
Time Frame: 24 weeks
Population: The Full Analysis Set 1 (FAS-1) consisted of all ICT naive randomized participants during the core phase.
Measure: Mean (95% Confidence Interval); unit: percentage of compliance
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 54 | 54
percentage of compliance | 89.45 [85.29 to 93.61] | 91.78 [87.81 to 95.75]
Statistical Analysis 1: Comparison: DFX DT vs DFX Granule; Test type: Superiority; p = 0.3598, ANCOVA; Least squares mean = 2.58, 95% CI 2-sided [-2.99 to 8.15], Standard Error of Mean 2.803

2. Primary Outcome: Change From Baseline in Serum Ferritin (SF) for Both Study Drug Formulations in ICT naïve Participants During the Core Phase
Description: The analysis included the comparison of means between the two treatment arms of change from baseline after 24 weeks of treatment in serum ferritin in pediatric ICT naïve participants with iron overload. The endpoint was assessed at Week 25 visit.
Time Frame: From Baseline to Week 25
Population: The Full Analysis Set 1 (FAS-1) consisted of all ICT naive randomized participants during the core phase.
Measure: Mean (95% Confidence Interval); unit: μg/L
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 54 | 54
μg/L
  Baseline | 2063.7 [1807.17 to 2320.15] | 1955.5 [1712.57 to 2198.49]
  Week 25: number analyzed (Participants) | 38 | 44
  Week 25 | 2216.3 [1929.59 to 2502.93] | 2228.4 [2011.69 to 2445.18]
  Change from Baseline to Week 25: number analyzed (Participants) | 38 | 44
  Change from Baseline to Week 25 | 250.5 [-84.63 to 585.58] | 340.0 [115.48 to 564.59]
Statistical Analysis 1: Comparison: DFX DT vs DFX Granule; Test type: Superiority; p = 0.2546, ANCOVA; Least squares mean = 176.36, 95% CI 2-sided [-129.00 to 481.72], Standard Error of Mean 153.933

3. Secondary Outcome: Percentage of Overall Compliance Using Stick Pack or Tablet Counts in ICT-naïve Participants During the Core Phase
Description: Compliance was calculated as the ratio of total count consumed to total count prescribed of deferasirox granule stick packs or dispersible tablets over 48 weeks of treatment.
Time Frame: 48 weeks
Population: The Full Analysis Set 1 (FAS-1) consisted of all ICT naive randomized participants during the core phase.
Measure: Mean (95% Confidence Interval); unit: percentage of compliance
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 54 | 54
percentage of compliance | 91.57 [87.65 to 95.49] | 94.80 [91.48 to 98.13]

4. Secondary Outcome: Change From Baseline in Serum Ferritin (SF) for Both Study Drug Formulations in ICT naïve Participants During the Core Phase
Description: The analysis included the comparison of means between the two treatment arms of change from baseline after 48 weeks of treatment in serum ferritin in pediatric ICT naïve participants with iron overload.
Time Frame: From Baseline to 48 weeks
Population: The Full Analysis Set 1 (FAS-1) consisted of all ICT naive randomized participants during the core phase.
Measure: Mean (95% Confidence Interval); unit: μg/L
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 54 | 54
μg/L | 305.8 [4.28 to 607.24] | 317.0 [69.10 to 564.88]

5. Secondary Outcome: Change From Baseline in Serum Ferritin (SF) for Both Study Drug Formulations in Pre-treated Participants During the Core Phase
Description: The analysis included the comparison of means between the two treatment arms of change from baseline after 25 weeks and after 48 weeks of treatment in serum ferritin in pre-treated participants. The analyses were performed at Week 25 and Week 48.
Time Frame: From Baseline to Week 25 and Week 48
Population: The Full Analysis Set 2 (FAS-2) consisted of all ICT pre-treated randomized participants during the core phase.
Measure: Mean (95% Confidence Interval); unit: μg/L
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 58 | 58
μg/L
  Change from Baseline to Week 25: number analyzed (Participants) | 48 | 52
  Change from Baseline to Week 25 | 59.0 [-210.88 to 328.79] | 150.3 [-59.43 to 360.01]
  Change from Baseline to Week 48: number analyzed (Participants) | 52 | 50
  Change from Baseline to Week 48 | 207.7 [-94.29 to 509.68] | 215.7 [-50.47 to 481.95]

6. Secondary Outcome: Change Over-time in Domain Score of Modified Satisfaction With Iron Chelation Therapy (mSICT) Using Patient Reported Outcomes (PRO) Questionnaires
Description: Participants aged between 10 years and less than 18 years at enrollment completed PRO questionnaires by themselves. The mSICT questionnaire for PRO consisted of 3 domains: adherence, satisfaction/preference, and concerns. The adherence domain had a minimum score of 6 and maximum score of 30; a lower score for adherence indicates better adherence. Satisfaction/preference domain had a minimum score of 2 and maximum score of 10; a lower score for satisfaction/preference indicates better satisfaction/preference. Concerns domain had a minimum score of 3 and maximum score of 15; a higher score for concerns indicate fewer concerns.
Time Frame: At Week 2, Week 3, Week 25 and Week 48
Population: The Full Analysis Set 3 (FAS-3) consisted of all randomized participants during the core phase. This includes only the participants aged between 10 years and less than 18 years with a valid assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 16 | 17
score on a scale
  Adherence (Week 2): number analyzed (Participants) | 13 | 15
  Adherence (Week 2) | 9.5 (2.30) | 7.6 (1.99)
  Adherence (Week 3) | 10.9 (4.95) | 6.6 (0.79)
  Adherence (Week 25): number analyzed (Participants) | 13 | 11
  Adherence (Week 25) | 11.9 (3.93) | 9.2 (3.31)
  Adherence (Week 48): number analyzed (Participants) | 13 | 15
  Adherence (Week 48) | 12.9 (4.17) | 8.4 (2.29)
  Satisfaction/preference (Week 2): number analyzed (Participants) | 13 | 15
  Satisfaction/preference (Week 2) | 5.2 (2.09) | 2.9 (1.36)
  Satisfaction/preference (Week 3) | 4.0 (1.32) | 3.1 (1.22)
  Satisfaction/preference (Week 25): number analyzed (Participants) | 13 | 11
  Satisfaction/preference (Week 25) | 5.5 (2.37) | 3.0 (1.10)
  Satisfaction/preference (Week 48): number analyzed (Participants) | 13 | 15
  Satisfaction/preference (Week 48) | 4.8 (2.24) | 3.1 (0.92)
  Concerns (Week 2): number analyzed (Participants) | 13 | 15
  Concerns (Week 2) | 13.1 (2.18) | 14.5 (1.06)
  Concerns (Week 3) | 13.4 (2.10) | 14.4 (0.80)
  Concerns (Week 25): number analyzed (Participants) | 13 | 11
  Concerns (Week 25) | 11.5 (3.13) | 14.5 (1.21)
  Concerns (Week 48): number analyzed (Participants) | 13 | 15
  Concerns (Week 48) | 12.8 (2.20) | 13.5 (2.75)

7. Secondary Outcome: Change Over-time in Domain Score of Modified Satisfaction With Iron Chelation Therapy (mSICT) Using Observer Reported Outcomes (ObsRO) Questionnaire (Caregiver's Perspective)
Description: The ObsRO questionnaires for participants aged between 2 years and less than 10 years were designed as observations made by caregivers such as the parent or legal guardian. The caregivers continued completing the ObsRO questionnaires even after the participant turned 10 years for consistency in responses. The mSICT questionnaire consisted of 2 domains: adherence and concerns per caregiver's perspective. The adherence domain had a minimum score of 5 and a maximum score of 25; a lower score for adherence indicates better adherence. The concerns domain had a minimum score of 1 and a maximum score of 5; a higher score for concerns indicates fewer concerns.
Time Frame: At Week 2, Week 3, Week 25 and Week 48
Population: The Full Analysis Set 3 (FAS-3) consisted of all randomized participants during the core phase. This includes only the participants aged between 2 years and less than 10 years with a valid assessment for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 73 | 74
score on a scale
  Adherence (Week 2): number analyzed (Participants) | 68 | 64
  Adherence (Week 2) | 7.7 (2.84) | 5.8 (1.32)
  Adherence (Week 3) | 7.8 (2.64) | 5.8 (1.43)
  Adherence (Week 25): number analyzed (Participants) | 61 | 53
  Adherence (Week 25) | 7.1 (2.35) | 6.5 (1.69)
  Adherence (Week 48): number analyzed (Participants) | 60 | 54
  Adherence (Week 48) | 7.5 (2.53) | 6.8 (2.57)
  Concerns (Week 2): number analyzed (Participants) | 68 | 64
  Concerns (Week 2) | 3.9 (1.32) | 4.5 (0.94)
  Concerns (Week 3) | 4.1 (1.31) | 4.7 (0.71)
  Concerns (Week 25): number analyzed (Participants) | 61 | 53
  Concerns (Week 25) | 4.3 (1.00) | 4.5 (0.89)
  Concerns (Week 48): number analyzed (Participants) | 60 | 54
  Concerns (Week 48) | 4.0 (1.24) | 4.6 (0.77)

8. Secondary Outcome: Change Over-time in Domain Score of Modified Satisfaction With Iron Chelation Therapy (mSICT) Using Observer Reported Outcomes (ObsRO) Questionnaire (Child's Perspective)
Description: The ObsRO questionnaires for participants aged between 2 years and less than 10 years were designed as observations made by caregivers such as the parent or legal guardian. The caregivers continued completing the ObsRO questionnaires even after the participant turned 10 years for consistency in responses. The mSICT questionnaire is presented for 2 domains: adherence and concerns per child's perspective. The adherence domain had a minimum score of 6 and a maximum score of 30; a lower score for adherence indicates better adherence. The concerns domain had a minimum score of 2 and a maximum score of 10; a higher score for concerns indicates fewer concerns.
Time Frame: At Week 2, Week 3, Week 25 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 73 | 74
score on a scale
  Adherence (Week 2): number analyzed (Participants) | 68 | 64
  Adherence (Week 2) | 12.1 (4.57) | 8.2 (2.28)
  Adherence (Week 3) | 11.7 (3.78) | 8.2 (2.64)
  Adherence (Week 25): number analyzed (Participants) | 61 | 53
  Adherence (Week 25) | 11.1 (3.82) | 9.1 (2.64)
  Adherence (Week 48): number analyzed (Participants) | 60 | 54
  Adherence (Week 48) | 11.3 (3.99) | 9.1 (3.00)
  Concerns (Week 2): number analyzed (Participants) | 68 | 64
  Concerns (Week 2) | 8.5 (2.29) | 9.2 (1.66)
  Concerns (Week 3) | 8.7 (2.00) | 8.8 (2.04)
  Concerns (Week 25): number analyzed (Participants) | 61 | 53
  Concerns (Week 25) | 8.6 (1.94) | 8.7 (1.85)
  Concerns (Week 48): number analyzed (Participants) | 60 | 54
  Concerns (Week 48) | 8.8 (1.75) | 9.0 (1.82)

9. Secondary Outcome: Change Over-time in Domain Score of Palatability Using Patient Reported Outcomes (PRO) Questionnaires
Description: The palatability questionnaire was used to measure: taste, aftertaste, whether medication was taken and how the participant perceived the amount of medication taken. This questionnaire had a minimum score of 0 and maximum score of 11; a higher score means better palatability. Participants aged between 10 years and less than 18 years at enrollment completed the PRO questionnaire by themselves.
Time Frame: At Week 2, Week 3, Week 25 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 16 | 17
score on a scale
  Week 2: number analyzed (Participants) | 13 | 15
  Week 2 | 8.8 (3.32) | 10.3 (1.91)
  Week 3 | 9.6 (2.83) | 10.9 (0.24)
  Week 25: number analyzed (Participants) | 13 | 11
  Week 25 | 9.2 (2.70) | 10.4 (1.80)
  Week 48: number analyzed (Participants) | 13 | 14
  Week 48 | 9.4 (3.07) | 11.0 (0.00)

10. Secondary Outcome: Change Over-time in Domain Score of Palatability Using Observer Reported Outcomes (ObsRO) Questionnaire
Description: The palatability questionnaire was used to measure: taste, aftertaste, whether medication was taken and how the participant perceived the amount of medication taken. This questionnaire had a minimum score of 0 and maximum score of 11; a higher score means better palatability. The ObsRO questionnaires for participants aged between 2 years and less than 10 years were designed as observations made by caregivers such as the parent or legal guardian. The caregivers continued completing the ObsRO questionnaires even after the participant turned 10 years for consistency in responses.
Time Frame: At Week 2, Week 3, Week 25 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 72 | 72
score on a scale
  Week 2: number analyzed (Participants) | 68 | 62
  Week 2 | 8.9 (3.13) | 10.9 (0.90)
  Week 3 | 9.4 (2.88) | 10.8 (0.79)
  Week 25: number analyzed (Participants) | 61 | 52
  Week 25 | 9.3 (2.83) | 10.6 (1.73)
  Week 48: number analyzed (Participants) | 60 | 53
  Week 48 | 9.0 (3.11) | 10.9 (0.96)

11. Secondary Outcome: Change Over Time in Weekly Dose Violation Rate Using Compliance Patient Reported Outcomes (PRO) Questionnaire
Description: The compliance questionnaire consisted of 2 items: 1. To assess if the medication was taken (yes/no) and 2. To record of the time when the medication was taken (with a not applicable option for participants who did not take their medication). Daily diary records were used to calculate the rate of dose violation in each study arm (doses missed completely or not taken before 12 PM). The dose violation rate was calculated as:
  [Number of dose violations / Drug exposure (days)] *100. Higher values represent more dose violations.
Time Frame: At Week 1, Week 13, Week 25, Week 37 and Week 48
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: percentage of days with dose violations
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 16 | 16
percentage of days with dose violations
  Week 1 | 26.86 (37.966) | 26.79 (38.992)
  Week 13: number analyzed (Participants) | 15 | 12
  Week 13 | 12.78 (31.000) | 23.41 (35.906)
  Week 25: number analyzed (Participants) | 12 | 9
  Week 25 | 13.19 (29.614) | 25.93 (42.583)
  Week 37: number analyzed (Participants) | 9 | 9
  Week 37 | 18.89 (32.745) | 30.16 (41.921)
  Week 48: number analyzed (Participants) | 7 | 6
  Week 48 | 2.86 (7.559) | 52.38 (52.424)

12. Secondary Outcome: Change Over Time in Weekly Dose Violation Rate Using Compliance Observer Reported Outcomes (ObsRO) Questionnaire
Description: The compliance questionnaire consisted of 2 items: 1. To assess if the medication was taken (yes/no) and 2. To record the time when the medication was taken (with a not applicable option for participants who did not take their medication). Daily diary records were used to calculate the rate of dose violation in each treatment arm (doses missed completely or not taken before 12 PM). The ObsRO questionnaires for participants aged between 2 years and less than 10 years were designed as observations made by caregivers such as the parent or legal guardian. The caregivers continued completing the ObsRO questionnaires even after the participant turned 10 years for consistency in responses. The dose violation rate was calculated as: [Number of dose violations / Drug exposure (days)] *100.
  Higher values represent more dose violations.
Time Frame: At Week 1, Week 13, Week 25, Week 37 and Week 48
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: percentage of days with dose violations
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 62 | 60
percentage of days with dose violations
  Week 1 | 18.80 (29.912) | 27.79 (37.577)
  Week 13: number analyzed (Participants) | 60 | 57
  Week 13 | 10.38 (27.374) | 18.65 (35.513)
  Week 25: number analyzed (Participants) | 48 | 53
  Week 25 | 7.79 (23.025) | 13.72 (31.813)
  Week 37: number analyzed (Participants) | 54 | 53
  Week 37 | 13.86 (31.769) | 20.01 (37.632)
  Week 48: number analyzed (Participants) | 36 | 34
  Week 48 | 13.56 (32.211) | 14.50 (31.123)

13. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the Core Phase
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation participant after providing written informed consent for participation in the study.
Time Frame: From Baseline to 48 weeks
Population: The Safety Set consisted of all participants who received at least 1 dose of study drug during the core phase. Three participants did not receive the study drug and hence were excluded from the safety set.
Measure: Count of Participants; unit: Participants
Groups:
- DFX DT - Core Phase: Participants received deferasirox (DFX) dispersible tablets (DT) orally once daily based on body weight for 48 weeks in the Core phase. The starting dose was 20mg/kg/day which was then adjusted based on tolerability, safety and efficacy considerations.
- DFX Granule - Core Phase: Participants received deferasirox (DFX) granules orally once daily based on body weight in the form of stick packs for 48 weeks in the Core phase. The starting dose was 14 mg/kg/day which was then adjusted based on tolerability, safety and efficacy considerations.
Arm/Group | DFX DT - Core Phase | DFX Granule - Core Phase
Number analyzed (Participants) | 111 | 110
Participants
  All AEs | 108 | 100
  All SAEs | 23 | 27

14. Secondary Outcome: Pre-dose Concentrations of Deferasirox to Support the Assessment of Compliance
Description: Pre-dose pharmacokinetic (PK) data from participants in the Pharmacokinetic Analysis Set 1 (PAS-1) were analyzed to assess variability of individual participant's compliance. A linear mixed effect power model to pre-dose samples which fulfill compliance criteria in terms of steady state (4 consecutive same doses prior to the PK sample drawn), time-windows (PK sample drawn 20 to 28 hours after previous dose) and without any vomiting episodes within the 4 hours prior to the PK sample were fitted. The model considered dose, treatment group, stratification factors and potential other factors, such as body weight as covariates.
Time Frame: At Weeks 1, 3, 5, 9, 13, 17, 21, 25, 29, 33, 37, 41, and 45
Population: Pharmacokinetic Analysis Set 1 (PAS-1) consisted of all participants who had at least one evaluable pre- or 3 hours post-dose PK concentration of deferasirox. The analysis included participants only with evaluable values.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/L
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 106 | 105
μmol/L
  Week 1: number analyzed (Participants) | 95 | 93
  Week 1 | 2.93 (369.5) | 1.40 (235.4)
  Week 3: number analyzed (Participants) | 59 | 73
  Week 3 | 14.2 (137.0) | 11.8 (117.1)
  Week 5: number analyzed (Participants) | 69 | 73
  Week 5 | 14.4 (115.7) | 11.7 (127.5)
  Week 9: number analyzed (Participants) | 68 | 74
  Week 9 | 20.1 (115.8) | 12.1 (97.1)
  Week 13: number analyzed (Participants) | 63 | 66
  Week 13 | 19.7 (124.2) | 13.5 (107.5)
  Week 17: number analyzed (Participants) | 62 | 56
  Week 17 | 18.4 (109.4) | 13.1 (135.3)
  Week 21: number analyzed (Participants) | 64 | 64
  Week 21 | 19.6 (120.4) | 13.4 (163.6)
  Week 25: number analyzed (Participants) | 60 | 62
  Week 25 | 17.1 (147.2) | 15.9 (108.6)
  Week 29: number analyzed (Participants) | 63 | 65
  Week 29 | 23.8 (111.3) | 13.2 (156.6)
  Week 33: number analyzed (Participants) | 65 | 69
  Week 33 | 21.4 (184.0) | 14.1 (175.6)
  Week 37: number analyzed (Participants) | 62 | 72
  Week 37 | 20.8 (137.1) | 14.6 (135.3)
  Week 41: number analyzed (Participants) | 66 | 71
  Week 41 | 21.8 (131.6) | 15.5 (134.7)
  Week 45: number analyzed (Participants) | 63 | 71
  Week 45 | 28.3 (141.2) | 19.0 (117.0)

15. Secondary Outcome: Concentrations of Deferasirox Between 2 and 4 Hours Post-dose at Weeks 5 and 9
Description: Post-dose pharmacokinetic (PK) data from participants in the Pharmacokinetic Analysis Set 1 (PAS-1) were analyzed along with Pre-dose PK data.
Time Frame: At Week 5 and Week 9
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μmol/L
Arm/Group | DFX DT | DFX Granule
Number analyzed (Participants) | 106 | 105
μmol/L
  Week 5 (3 hour post-dose): number analyzed (Participants) | 66 | 70
  Week 5 (3 hour post-dose) | 65.2 (80.5) | 53.2 (86.2)
  Week 9 (3 hour post-dose): number analyzed (Participants) | 62 | 61
  Week 9 (3 hour post-dose) | 70.4 (77.0) | 59.8 (61.7)

16. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) During the Entire Granule Period
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation after participant providing written informed consent for participation in the study. In the DFX Granules arm, AEs are reported since the initial randomization to the arm in the core phase and continuing in the extension phase. In the DFX cross-over arm, AEs are reported for participants since the participant crossed-over from dispersible tablet to granules in the extension phase only.
Time Frame: From Baseline to 305 weeks
Population: The Safety Set consisted of all participants who received at least 1 dose of granule formulation during the core or extension phase. The participants in the extension phase received granules regardless of which arm they were initially randomized.
Measure: Count of Participants; unit: Participants
Groups:
- DFX DT Cross-over Granule - Optional Extension Phase: After the Core phase, participants could enter the Optional Extension phase and cross over to DFX granules administered orally once daily in the form of stick packs for up to 5 years. Participants entering the Optional Extension phase received the equivalent strength-adjusted DFX granules dose corresponding to the last DT dose in the Core phase taking dose adjustment guidelines into account.
- DFX Granules - Core and Optional Extension Phase: Participants received deferasirox (DFX) granules orally once daily based on body weight in the form of stick packs for 48 weeks in the Core phase. The starting dose was 14 mg/kg/day which was then adjusted based on tolerability, safety and efficacy considerations. After the Core phase, participants could enter the Optional Extension phase and continued receiving DFX granules at the same dose as was given at the end of the Core phase taking dose adjustment guidelines into account for up to 5 years.
Arm/Group | DFX DT Cross-over Granule - Optional Extension Phase | DFX Granules - Core and Optional Extension Phase
Number analyzed (Participants) | 69 | 110
Participants
  AEs | 64 | 106
  Suspected AEs | 48 | 73
  SAEs | 22 | 38
  Suspected SAEs | 4 | 7

17. Secondary Outcome: Number of Participants With Adverse Events of Special Interest (AESI) During the Entire Granule Period
Description: An adverse event (AE) is any untoward medical occurrence (e.g. any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a clinical investigation after participant providing written informed consent for participation in the study. In the DFX Granules arm, AEs are reported since the initial randomization to the arm in the core phase and continuing in the extension phase. In the DFX cross-over arm, AEs are reported for participants since the participant crossed-over from dispersible tablet to granules in the extension phase only. AESI included active monitoring for renal toxicity; including renal failure, hepatic toxicity; including hepatic failure, and gastrointestinal hemorrhage
Time Frame: From Baseline to 305 weeks
Population: as for outcome 16
Measure: Count of Participants; unit: Participants
Arm/Group | DFX DT Cross-over Granule - Optional Extension Phase | DFX Granules - Core and Optional Extension Phase
Number analyzed (Participants) | 69 | 110
Participants
  Any AESI | 52 | 79
  Gastrointestinal hemorrhages | 3 | 4
  Hearing loss | 5 | 5
  Lens opacities, Retinal changes and Optic neuritis | 0 | 2
  Liver disorders - Hepatic failure | 1 | 0
  Liver disorders - Increased liver transaminases | 16 | 46
  Peripheral blood cytopenias | 5 | 7
  Renal disorders - Acute renal failure | 1 | 0
  Renal disorders - Increased serum creatinine | 4 | 8
  Renal disorders -Proteinuria | 40 | 49
  Renal disorders - Renal tubular disorders | 4 | 0
  Severe Cutaneous Adverse Reactions (SCARs) | 0 | 1

18. Other Pre Specified Outcome: Exposure-Response Relationship in Relation to Pre- and Post-Dose Deferasirox Concentrations (PK/PD Relationship)
Description: This outcome measure explores exposure-response relationships for measures of safety and effectiveness through serum creatinine change from baseline, notable serum creatinine values, serum creatinine clearance change form baseline and notable serum creatinine clearance categories, serum ferritin change from baseline, in relationship to derived PK parameters for pre- and post-dose deferasirox concentrations.
Time Frame: From Baseline to 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From initial randomization up to 48 weeks (Core phase) and Up to 5 years from entering the extension phase (Optional Extension phase)
Description: The Safety Set consisted of all participants who received at least 1 dose of granule formulation during the core or extension phase. The participants in extension phase received granules regardless of which arm they were initially randomized. Three participants did not receive the study drug and hence were excluded from the safety set.
Groups:
- DFX DT- Core Phase: Participants received deferasirox (DFX) dispersible tablets (DT) orally once daily based on body weight for 48 weeks in the Core phase. The starting dose was 20mg/kg/day which was then adjusted based on tolerability, safety and efficacy considerations.
- DFX Granules - Core Phase: Participants received deferasirox (DFX) granules orally once daily based on body weight in the form of stick packs for 48 weeks in the Core phase. The starting dose was 14 mg/kg/day which was then adjusted based on tolerability, safety and efficacy considerations.
- DFX Granules - Optional Extension Phase: After the Core phase, participants could enter the Optional Extension phase and continued receiving DFX granules at the same dose as was given at the end of the Core phase taking dose adjustment guidelines into account for up to 5 years.
Arm/Group | DFX DT- Core Phase | DFX DT Cross-over Granule - Optional Extension Phase | DFX Granules - Core Phase | DFX Granules - Optional Extension Phase
All-Cause Mortality (participants affected / at risk) | 0/111 | 1/69 | 0/110 | 0/77
Serious Adverse Events (participants affected / at risk) | 23/111 | 22/69 | 27/110 | 20/77
Other Adverse Events (participants affected / at risk) | 104/111 | 63/69 | 97/110 | 63/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DFX DT- Core Phase (N=111) | DFX DT Cross-over Granule - Optional Extension Phase (N=69) | DFX Granules - Core Phase (N=110) | DFX Granules - Optional Extension Phase (N=77)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Hypersplenism (Blood and lymphatic system disorders) | 1 | 0 | 0 | 1
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Sickle cell anaemia with crisis (Blood and lymphatic system disorders) | 5 | 0 | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Malpositioned teeth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Stress ulcer (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 4 | 1 | 4 | 2
Sudden death (General disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0 | 3
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Amoebiasis (Infections and infestations) | 1 | 0 | 0 | 0
Ascariasis (Infections and infestations) | 1 | 0 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 0 | 1 | 0
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 0 | 0 | 2 | 0
Bronchitis (Infections and infestations) | 3 | 0 | 0 | 1
Bronchitis viral (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Dengue fever (Infections and infestations) | 1 | 1 | 2 | 1
Dengue haemorrhagic fever (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 4 | 2 | 4
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis salmonella (Infections and infestations) | 0 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0
Otitis media acute (Infections and infestations) | 1 | 0 | 1 | 0
Parotid abscess (Infections and infestations) | 0 | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 0 | 1 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 2 | 0 | 1
Pharyngotonsillitis (Infections and infestations) | 0 | 0 | 1 | 1
Pneumonia (Infections and infestations) | 3 | 1 | 1 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 0 | 1 | 0
Scarlet fever (Infections and infestations) | 0 | 1 | 0 | 0
Shigella infection (Infections and infestations) | 1 | 0 | 0 | 0
Sinobronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 0
Subcutaneous abscess (Infections and infestations) | 0 | 1 | 0 | 0
Systemic viral infection (Infections and infestations) | 0 | 0 | 1 | 1
Tonsillitis (Infections and infestations) | 2 | 2 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Varicella (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 2 | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Wound infection (Infections and infestations) | 0 | 0 | 1 | 0
Craniofacial fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Lip injury (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 2 | 0 | 0
Urine protein/creatinine ratio increased (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 2 | 0 | 2
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Lactase deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tension headache (Nervous system disorders) | 0 | 0 | 0 | 1
Fanconi syndrome acquired (Renal and urinary disorders) | 1 | 3 | 0 | 0
Acute chest syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Obstructive sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Drug reaction with eosinophilia and systemic symptoms (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DFX DT- Core Phase (N=111) | DFX DT Cross-over Granule - Optional Extension Phase (N=69) | DFX Granules - Core Phase (N=110) | DFX Granules - Optional Extension Phase (N=77)
Abdominal pain (Gastrointestinal disorders) | 4 | 4 | 12 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 3 | 4 | 4
Constipation (Gastrointestinal disorders) | 5 | 4 | 2 | 0
Dental caries (Gastrointestinal disorders) | 7 | 3 | 5 | 2
Diarrhoea (Gastrointestinal disorders) | 14 | 7 | 9 | 6
Gastritis (Gastrointestinal disorders) | 0 | 4 | 1 | 4
Nausea (Gastrointestinal disorders) | 8 | 3 | 4 | 1
Vomiting (Gastrointestinal disorders) | 15 | 9 | 9 | 4
Pyrexia (General disorders) | 24 | 15 | 26 | 16
Bronchitis (Infections and infestations) | 4 | 4 | 3 | 3
COVID-19 (Infections and infestations) | 0 | 8 | 0 | 9
Gastroenteritis (Infections and infestations) | 8 | 5 | 5 | 6
Influenza (Infections and infestations) | 4 | 2 | 5 | 7
Nasopharyngitis (Infections and infestations) | 12 | 14 | 11 | 11
Pharyngitis (Infections and infestations) | 3 | 12 | 11 | 7
Rhinitis (Infections and infestations) | 3 | 3 | 9 | 1
Systemic viral infection (Infections and infestations) | 0 | 1 | 0 | 4
Tonsillitis (Infections and infestations) | 2 | 5 | 7 | 3
Upper respiratory tract infection (Infections and infestations) | 34 | 23 | 31 | 24
Urinary tract infection (Infections and infestations) | 2 | 6 | 3 | 6
Alanine aminotransferase increased (Investigations) | 15 | 11 | 20 | 11
Aspartate aminotransferase increased (Investigations) | 11 | 8 | 12 | 7
Bilirubin conjugated increased (Investigations) | 16 | 2 | 12 | 3
Blood bilirubin increased (Investigations) | 4 | 4 | 3 | 5
Blood creatinine increased (Investigations) | 3 | 3 | 0 | 6
Transaminases increased (Investigations) | 7 | 2 | 9 | 8
Urine protein/creatinine ratio increased (Investigations) | 39 | 36 | 27 | 28
Headache (Nervous system disorders) | 8 | 5 | 9 | 2
Proteinuria (Renal and urinary disorders) | 8 | 4 | 9 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 14 | 15 | 9
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 8 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 5 | 5
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 7 | 6
Rash (Skin and subcutaneous tissue disorders) | 7 | 2 | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-06-24): https://cdn.clinicaltrials.gov/large-docs/12/NCT02435212/Prot_000.pdf
  • Statistical Analysis Plan (2024-02-21): https://cdn.clinicaltrials.gov/large-docs/12/NCT02435212/SAP_001.pdf